CLINICAL TRIAL: NCT01470690
Title: Pharmacokinetic Study of the HCV Protease Inhibitor Bo-cePRevir and the Proton Pump Inhibitor OMeprazOle (PROMO)
Acronym: PROMO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UMCN-AKF 10.06
Record Dates: First submitted 2011-11-01; First posted 2011-11-11 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: HCV Infections; Gastric Acid-related Disorders
Keywords: HVC infection; gastric acid-related disorders; proton pump inhibitor; interaction; pharmacokinetics; boceprevir; omeprazole
MeSH Terms: interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- boceprevir (Active Comparator): Boceprevir 800 mg TID for 4 consecutive days + a single dose of 800 mg on Day 5 (BOC alone)
  Interventions: Drug: boceprevir
- omeprazole (Active Comparator): Omeprazole 40 mg QD for 5 consecutive days (OME alone)
  Interventions: Drug: Omeprazole
- boceprevir+omeprazole (Experimental): Omeprazole 40 mg QD for 5 consecutive days combined with boceprevir 800 mg TID for 4 consecutive days + a single dose of 800 mg on Day 5 (BOC+OME)
  Interventions: Drug: boceprevir; Drug: Omeprazole

INTERVENTIONS:
Drug: boceprevir — Boceprevir 800 mg TID for 4 consecutive days + a single dose of 800 mg on Day 5
  Arms: boceprevir; boceprevir+omeprazole
Drug: Omeprazole — Omeprazole 40 mg QD for 5 consecutive days
  Arms: boceprevir+omeprazole; omeprazole

SUMMARY:
The objective of this study is to determine the effect of multiple dose omeprazole on the pharmacokinetics of boceprevir and vice versa.

Furthermore, the safety of steady state boceprevir combined with multiple dose omeprazole will be evaluated.

DETAILED DESCRIPTION:
It is known that some drugs can significantly influence the bioavailability of other drugs. For example the proton pump inhibitors decrease the absorption of some protease inhibitors used in HIV treatment or of some oral tyrosine kinase inhibitors used in oncology. Proton pump inhibitors increase the pH in the stomach and might therefore decrease the solubility of other drugs with decreased absorption as a consequence.

Boceprevir (BOC) is an Hepatitis C (HCV) NS3 serine protease inhibitor that has recently received FDA approval for the treatment of chronic HCV infection. The drug substance is slightly soluble in water and administration with food increases the oral bioavailability of BOC relative to the fasted state, by 40% to 60% based on AUC.

Omeprazole (OME) is the most frequently used proton pump inhibitor. It is the second most prescribed drug in The Netherlands, with 5 million prescriptions a year.

OME is metabolized by CYP2C19 and CYP3A4 and is known to induce CYP1A2 and inhibit CYP2C19. BOC is a potent inhibitor of CYP3A4/5 and is not metabolised by CYP1A2 or CYP2C19. No interaction on metabolism of BOC is expected. However, an increase of OME levels may be expected due to the inhibition of CYP3A4 by BOC.

As proton pump inhibitors are widely used it is relevant to know if a drug-drug interaction between proton pump inhibitors and BOC exists which might influence the bioavailability of BOC.

This study is designed to determine the effect of multiple dose omeprazole on the pharmacokinetics of boceprevir and vice versa.

Furthermore, the safety of steady state boceprevir combined with multiple dose omeprazole will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 and not older than 55 years at screening.
* Subject does not smoke more than 10 cigarettes, 2 cigars, or 2 pipes per day for at least 3 months prior to the first dosing.
* Subject has a Quetelet Index (Body Mass Index) of 18 to 30 kg/m2, extremes included.
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* Subject is in good age-appropriate health condition as established by medical history, physical examination, electrocardiography, results of biochemistry, haematology and urinalysis testing within 4 weeks prior to Day 1.

Results of biochemistry, haematology and urinalysis testing should be within the laboratory's reference ranges. If laboratory results are not within the reference ranges, the subject is included on condition that the Investigator judges that the deviations are not clinically relevant. This should be clearly recorded.

* Subject has a normal blood pressure and pulse rate, according to the Investigator's judgement.

Exclusion Criteria:

* Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
* Positive HIV test.
* Positive hepatitis B or C test.
* Pregnant female (as confirmed by an HCG test performed less than 4 weeks before Day 1) or breastfeeding female. Female subjects of childbearing potential without adequate contraception, e.g. hysterectomy, bilateral tubal ligation, (non-hormonal) intrauterine device, total abstinence, double barrier methods, or two years post-menopausal. They must agree to take precautions in order to prevent a pregnancy throughout the entire conduct of the trial.
* Therapy with any drug (for two weeks preceding dosing), except for paracetamol.
* Relevant history or presence of pulmonary disorders (especially COPD), cardiovascular disorders, neurological disorders (especially seizures and migraine), psychiatric disorders, gastro-intestinal disorders, renal and hepatic disorders, hormonal dis-orders (especially diabetes mellitus), coagulation disorders.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* History of or current abuse of drugs, alcohol or solvents.
* Inability to understand the nature and extent of the trial and the procedures required.
* Participation in a drug trial within 60 days prior to the first dose.
* Donation of blood within 60 days prior to the first dose.
* Febrile illness within 3 days before Day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
boceprevir concentrations | AUC: pre-dose, 0.5, 1. 1.5, 2, 2.5, 3, 4, 5, 6 and 8h
  to determine the effect of chronic use of omeprazole on the steady state pharmacokinetics of boceprevir

SECONDARY OUTCOMES:
omeprazole concentrations | AUC: pre-dose, 0.5, 1. 1.5, 2, 2.5, 3, 4, 5, 6 and 8h
  to determine the effect of chronic use of boceprevir on the steady state pharmacokinetics of omeprazole
adverse events | entire study
  to determine the safety of combined use of boceprevir and omeprazole

CONTACTS AND LOCATIONS:
Overall Officials: David Burger, Prof PharmD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Crcn, Runmc, Nijmegen, Netherlands

REFERENCES:
- [Result] de Kanter CT, Colbers AP, Blonk MI, Verweij-van Wissen CP, Schouwenberg BJ, Drenth JP, Burger DM. Lack of a clinically significant drug-drug interaction in healthy volunteers between the HCV protease inhibitor boceprevir and the proton pump inhibitor omeprazole. J Antimicrob Chemother. 2013 Jun;68(6):1415-22. doi: 10.1093/jac/dkt032. Epub 2013 Feb 20. PMID 23429642
- See also: Link to abstract on AASLD 2012 liver learning website, containing results of the PROMO study. — http://liverlearning.aasld.org/aasld/2012/thelivermeeting/24342/klaartje.de.kanter.influence.of.the.proton.pump.inhibitor.omeprazole.on.the.html?history_id=65835